CLINICAL TRIAL: NCT04284787
Title: BLockade of PD-1 Added to Standard Therapy to Target Measurable Residual Disease in Acute Myeloid Leukemia 2 (BLAST MRD AML-2): A Randomized Phase 2 Study of the Venetoclax, Azacitadine, and Pembrolizumab (VAP) Versus Venetoclax and Azacitadine as First Line Therapy in Older Patients With Acute Myeloid Leukemia (AML) Who Are Ineligible or Who Refuse Intensive Chemotherapy
Brief Title: BLAST MRD AML-2: BLockade of PD-1 Added to Standard Therapy to Target Measurable Residual Disease in Acute Myeloid Leukemia 2- A Randomized Phase 2 Study of Anti-PD-1 Pembrolizumab in Combination With Azacitidine and Venetoclax as Frontline Therapy in Unfit Patients With Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-01016; NCI-2020-01016 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2000031641; 10334 (Other: Yale University Cancer Center LAO); 10334 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2020-02-25; First posted 2020-02-26 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Acute Myeloid Leukemia Post Cytotoxic Therapy; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Biopsy; Specimen Handling; pembrolizumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (AZA, VEN) (Active Comparator): See Detailed Description
  Interventions: Drug: Azacitidine; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Venetoclax
- Arm II (AZA, VEN, pembrolizumab) (Experimental): See Detailed Description
  Interventions: Drug: Azacitidine; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Biological: Pembrolizumab; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood specimen collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
  Arms: Arm II (AZA, VEN, pembrolizumab)
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies how well azacitidine and venetoclax with or without pembrolizumab work in treating older patients with newly diagnosed acute myeloid leukemia. Chemotherapy drugs, such as azacitidine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving azacitidine and venetoclax with pembrolizumab may increase the rate of deeper/better responses and reduce the chance of the leukemia coming back in patients with newly diagnosed acute myeloid leukemia compared to conventional therapy of azacitidine and venetoclax alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the percentage of patients with minimal residual disease (MRD) negative complete remission (CR) (MRD-CR) or complete remission with incomplete count recovery (MRD-CRi) with azacitidine (AZA) + venetoclax (VEN) with pembrolizumab during the first 6 cycles and compare to control arm.

SECONDARY OBJECTIVES:

I. Assess the investigator-assessed rates of CR/CRi/partial remission (PR)/morphological leukemia free state (MLFS) as defined per the modified International Working Group (IWG) 2003 response criteria with AZA + VEN with pembrolizumab, as well as rates of MRD negative MLFS.

II. Rates of complete remission with partial count recovery (CRh) and hematologic improvement (HI) to red blood cells and platelets.

III. Assess time to MRD negativity and duration of MRD negative state, event free survival (EFS), relapse free survival (RFS), calculated as the time from initial treatment to either disease relapse or death, duration of response (DOR, defined as the time from first CR/CRi to the date of the first documented relapse or death, whichever occurs first) and overall survival (OS).

IV. Assess the proportion of patients who develop severe toxicity.

EXPLORATORY OBJECTIVES:

I. MRD assessment by duplex sequencing (DS) and comparing DS and multiparameter flow cytometry for MRD detection as an exploratory biomarker.

II. Assessment of immune-checkpoint expression and dynamic change of immune cell subsets in response to the combination of checkpoint-inhibition and backbone combination in acute myeloid leukemia (AML).

III. High-throughput sequencing of the T-cell receptor (TCR) Vb CDR3 regions on ﬂow cytometrically sorted t-cell subsets to assess the effect of immunotherapy on the diversity of the t-cell repertoire and assess for correlation to clinical outcomes.

IV. Investigation of protein signatures and ribonucleic acid (RNA) signatures associated with response and efficacy using O-link cytokine panel and RNA-sequencing (seq), respectively.

V. Determination of mutational load by whole exome sequencing to assess for correlation with clinical outcomes, immune infiltrating profile, and T cell repertoire diversity and clonality.

VI. Profiling of deoxyribonucleic acid (DNA) methylation patterns before and after treatment to assess for correlation to response to treatment.

VII. Correlate gut microbiome at baseline and changes in the microbiome with clinical response, both in standard chemotherapy and immunotherapy/chemotherapy therapy settings.

VIII. MRD assessment using duplex sequencing strategy for circulating cell-free tumor DNA and correlation with long-term outcomes.

IX. Exploring different thresholds of MRD negativity using flow cytometry aside from the 0.1% level that will be used for the primary endpoint purposes (e.g. 0.01%).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (AZA + VEN):

INDUCTION THERAPY PHASE: Patients receive azacitidine intravenously (IV) over 10-40 minutes or subcutaneously (SC) on days 1-7 or days 1-5 in week 1 and 1-2 in week 2. Patients also receive venetoclax orally (PO) on days 1-28 of cycle 1 and days 1-21 or 1-28 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY PHASE: Patients receive azacitidine IV over 10-40 minutes or SC on days 1-7 or days 1-5 in week 1 and 1-2 in week 2. Patients also receive venetoclax PO on days 1-21 or 1-28 (depending on count recovery) for all cycles. Cycles repeat every 28 days for up to 3 years in the absence of disease progression or unacceptable toxicity. After completion of 24 cycles, patients who respond to treatment or have stable disease (SD) may continue treatment per physician discretion.

ARM II (AZA + VEN + PEMBROLIZUMAB):

INDUCTION THERAPY PHASE: Patients receive pembrolizumab IV over 30 minutes on day 8 of cycle 1 and every 3 weeks in cycle 2-6, azacitidine IV over 10-40 minutes or SC on days 1-7 or days 1-5 in week 1 and 1-2 in week 2, and venetoclax PO on days 1-28 of cycle 1 and days 1-21 or 1-28 of subsequent cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY PHASE: Patients receive pembrolizumab IV over 30 minutes every 3 weeks, azacitidine IV over 10-40 minutes or SC on days 1-7 or days 1-5 in week 1 and 1-2 in week 2, and venetoclax PO on days 1-21 or 1-28 (depending on count recovery) for all cycles. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. After completion of 24 cycles, patients who respond to treatment or have SD may continue treatment with azacitidine and venetoclax per physician discretion.

Patients in both arms also undergo echocardiography (ECHO) or multigated acquisition (MUGA) scan during screening and bone marrow biopsy and/or aspiration and collection of blood samples throughout the trial, as well as a skin biopsy at baseline.

Patients are followed up every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and pathologically-confirmed, previously untreated AML as defined by World Health Organization (WHO) criteria. Bone marrow biopsy, or aspirate or peripheral blood that were obtained up to 3 weeks before signing consent are allowed for purposes of confirming AML diagnosis for eligibility purposes. Secondary AML arising from prior myelodysplastic syndrome (MDS), as long as they have not received more than full cycle of hypomethylating agent therapy for MDS, and therapy related (t)-AML are also allowed. AML arising from antecedent hematologic disorders defined as prior MDS, myeloproliferative neoplasm (MPN), or aplastic anemia are allowed. Note 1: Patients must have evidence of bone marrow involvement on aspirate or biopsy. Patients with only extramedullary disease and no bone marrow involvement will be excluded. Note 2: Every effort should be made to get an aspirate for central flow assessment at screening and all subsequent required time points, but in cases where an aspirate cannot be collected-including dry taps-the patient will not be excluded and assessments will be performed on peripheral blood (PB) which should be collected at every time that bone marrow (BM) is collected. Note 3: Some patients with AML require initiation of therapy quickly after diagnosis, and full metaphase karyotype results in some centers can take 2-3 weeks to result. To avoid this issue being an impediment to accrual to study or to cause delays in initiation of therapy in patients who need fast initiation of therapy, we allow use of karyotype and/or fluorescence in situ hybridization (FISH) results on samples from blood or marrow that were obtained up to 3 weeks before signing consent for purposes of eligibility and stratification. In any case, results from FISH or karyotype should exclude presence of core-binding factor (CBF) abnormalities by time of randomization
* Age >= 60 years
* Patients who are ineligible for intensive chemotherapy according to treating physician's assessment or who refuse intensive chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* Prior use of lenalidomide, erythropoiesis-stimulating agents (ESAs), and growth factors is allowed if used to treat prior MDS. AML must be previously untreated except for hydroxyurea, or all-trans retinoic acid (ATRA) for suspicion of APL but both should be discontinued prior to initiation of study therapy. Hypomethylating agents are not allowed to have been used for AML therapy. If hypomethylating agent therapy was used for prior MDS or MPN therapy then it should not have exceeded one full cycle. Note: One dose of prophylactic intrathecal therapy is allowed during or before screening if a lumbar puncture is performed to rule out central nervous system (CNS) involvement
* Hydroxyurea or leukopheresis are allowed for management of hyperleukocytosis, as well as ATRA, before initiation of study therapy. White blood cell (WBC) count must be < 25 x 10^9/L to start on study therapy per venetoclax label. Hydroxyurea and ATRA may be administered up to one day prior to start of study treatment
* Intermediate-risk or poor risk AML as well as favorable risk by National Comprehensive Cancer Network (NCCN)/European LeukemiaNet (ELN) with the exception of "good-risk" cytogenic profile (i.e., for eligibility patient should lack the presence of t(8;21), (inv[16] or t[16;16]), or t(15;17) by full cytogenetics or FISH). Clarification: We allow use of karyotype and/or FISH results (as well as FLT3 results) on samples from blood or marrow that were obtained up to 3 weeks before signing consent for purposes of eligibility and stratification. Adverse karyotype can be determined based on FISH results (e.g., loss of chromosome 7 or 5 or 3 or more abnormalities) based on the specific probes used in the FISH. If results of full metaphase karyotype are not available and the available FISH results do not suggest an adverse karyotype, and there is a need to initiate therapy before those full results are available, then the patient can be stratified into the unknown/intermediate NCCN cytogenetic group for randomization purposes. In any case, results from FISH or karyotype should show that core-binding factor (CBF) abnormalities are NOT present by at time of randomization as the presence of CBF abnormalities is an exclusion factor
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (CrCl) >= 60 mL/min for patient with creatinine levels > 1.5 x institutional ULN

  * Creatinine clearance (CrCl) should be calculated per institutional standard
  * Glomerular filtration rate (GFR) can also be used in place of creatinine or CrCl
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for patients with total bilirubin levels > 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN OR =< 5 x ULN for patients with liver metastases
* Patients who are human immunodeficiency virus (HIV) positive may participate IF they meet the following eligibility requirements:

  * They must be stable on their anti-retroviral regimen, and they must be healthy from an HIV perspective
  * Patients must have an undetectable HIV viral load
* Patients with a known history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients who have undergone major surgery must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months). Female patients of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication. Male patients who have a female partner of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. NOTE: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients with CBF-AML and acute promyelocytic leukemia (APL)
* Received a prior anti-cancer monoclonal antibodies (mAb) within 4 weeks prior to study registration or have not recovered (recovery defined as baseline or =< grade 1) from adverse events (AEs) due to agents administered more than 4 weeks earlier
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Patients who have had chemotherapy, targeted small molecule therapy (aside from imatinib, dasatinib, or nilotinib, hydroxyurea, or ATRA), or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Left ventricular ejection fraction < 50% as determined by either echocardiogram or MUGA
* Patients who have not recovered from AEs due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of =< grade 2 neuropathy and alopecia

  * NOTE: Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-CNS disease
* Patients currently participating and receiving study therapy or have participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment are ineligible
* History of hypersensitivity to pembrolizumab (MK-3475) or any of its excipients, or other agents used in this study
* Current use of systemic corticosteroids or immunosuppressive agents

  * EXCEPTION: Low doses of steroids (< 10 mg of prednisone or equivalent dose of other steroid), used for treatment of non-hematologic medical condition (e.g., chronic adrenal insufficiency) inhaled corticosteroids, or topical steroids are permitted
* Other active primary malignancy (other than non-melanomatous skin cancer or carcinoma in situ of the cervix) requiring treatment or limiting expected survival to =< 2 years

  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment (other than hormonal therapy for their cancer)
* Patient with known active CNS disease and/or carcinomatous meningitis before study enrollment. Assessment of the cerebrospinal fluid (CSF) is not required to enroll in the study unless there is clinical suspicion for CNS involvement. However, if CSF assessment is performed for any reason, there should be no evidence of active leukemia in the CSF as per investigator judgement. Up to one dose of prophylactic intrathecal chemotherapy is allowed prior to study enrollment. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of protocol treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to protocol treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Patients who received prior allogenic transplant
* Patient with a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Patient with a diagnosis of immunodeficiency or receiving high dose systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of treatment
* Patient with active autoimmune disease except for patients with hypothyroidism and vitiligo that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Patient with a known history of non-infectious pneumonitis that required the use of steroids or current non-infectious pneumonitis
* Patient with active uncontrolled infection
* Patient with a known history of active TB (Bacillus tuberculosis)
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because pembrolizumab (MK-3475) is humanized antibody with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab, breastfeeding should be discontinued if the mother is treated with pembrolizumab. These potential risks may also apply to other agents used in this study
* Patients with no bone marrow involvement (i.e., those with only extramedullary disease)
* Patients who received prior hypomethylating agent (HMA) therapy for more than one full cycle in treatment for prior MDS. Patient must not have received HMA therapy for treatment of AML
* Patients that received a live vaccine within 30 days of planned start of study therapy

  * NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist [registered trademark]) are live attenuated vaccines, and are not allowed
* Patients with active hemolytic anemia requiring immunosuppressive therapy or other pharmacologic treatment. Patients who have a positive Coombs test but no evidence of hemolysis are NOT excluded from participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2026-01-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amer M Zeidan, Principal Investigator — Yale University Cancer Center LAO
Locations (29):
- United States (29):
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (AZA, VEN): See Detailed Description
  Azacitidine: Given IV or SC
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood specimen collection
  Bone Marrow Aspiration: Undergo bone marrow aspiration
  Bone Marrow Biopsy: Undergo bone marrow biopsy
  Echocardiography: Undergo ECHO
  Multigated Acquisition Scan: Undergo MUGA scan
  Venetoclax: Given PO
- Arm II (AZA, VEN, Pembrolizumab): See Detailed Description
  Azacitidine: Given IV or SC
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo blood specimen collection
  Bone Marrow Aspiration: Undergo bone marrow aspiration
  Bone Marrow Biopsy: Undergo bone marrow biopsy
  Echocardiography: Undergo ECHO
  Multigated Acquisition Scan: Undergo MUGA scan
  Pembrolizumab: Given IV
  Venetoclax: Given PO
Period: Overall Study
Arm/Group | Arm I (AZA, VEN) | Arm II (AZA, VEN, Pembrolizumab)
Started | 31 | 29
Received Trial Therapy | 29 | 29
Completed Trial Therapy | 0 | 0
Completed (No participants completed trial therapy.) | 0 | 0
Not Completed | 31 | 29
Not completed — Disease Progression | 9 | 12
Not completed — Physician Decision | 12 | 7
Not completed — Transplant | 5 | 4
Not completed — Death | 1 | 2
Not completed — Adverse Event | 0 | 4
Not completed — Non-adherence | 2 | 0
Not completed — Lack of Efficacy | 2 | 0

BASELINE CHARACTERISTICS:
Population: Those receiving treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (AZA, VEN) | Arm II (AZA, VEN, Pembrolizumab) | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Median (Full Range); unit: years] | 73 [62 to 79] | 74 [63 to 82] | 73.5 [62 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 18 | 20 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 24 | 24 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58
ECOG PS [Count of Participants; unit: Participants] — The ECOG Performance Status Scale describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). It ranges from 0 (fully functional) to 5 (dead). https://ecog-acrin.org/resources/ecog-performance-status/
  Participants
    0 | 6 | 7 | 13
    1 | 19 | 13 | 32
    2 | 4 | 7 | 11
    MISSING | 0 | 2 | 2
ELN 2022 risk [Count of Participants; unit: Participants] — The 2022 European LeukemiaNet (ELN) AML is a risk stratification system.
  Participants
    Favorable | 4 | 5 | 9
    Intermediate | 5 | 4 | 9
    Adverse | 20 | 20 | 40
Clinically Relevant Mutations [Count of Participants; unit: Participants]
  TP53 | 4 | 5 | 9
  NPM1 | 4 | 5 | 9
  KRAS/NRAS | 4 | 7 | 11
  FLT3 | 1 | 4 | 5
  Secondary ontogeny | 16 | 15 | 31
  Missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Minimal Residual Disease Negative Complete Remission (MRD-CR) or MRD-complete Remission With Incomplete Count Recovery (Cri) With Azacitidine (AZA) + Venetoclax (VEN) With MK-3475 (Pembrolizumab)
Time Frame: Up to 6 cycles (each cycle is 28 days)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (AZA, VEN) | Arm II (AZA, VEN, Pembrolizumab)
Number analyzed (Participants) | 29 | 29
Participants
  MRD-negative CR/CRi | 13 | 13
  MRD-negative CR | 7 | 7
  No MRD-negative CR/CRi or lack thereof | 9 | 9

2. Secondary Outcome: Proportion of Patients Who Develop Severe Toxicity
Time Frame: Up to cycle 2 (each cycle is 28 days)
Population: the first 6 participants were assessed for severe pembrolizumab related toxicity, 1 participant was not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm II (AZA, VEN, Pembrolizumab)
Number analyzed (Participants) | 5
Participants | 0

3. Other Pre Specified Outcome: Biomarkers or Serial Measurements of Biomarkers Associated With Response Outcomes
Description: A univariate logistic regression will be selected to assess baseline biomarkers associated with response outcomes. The dynamic changes of PD-L1/ PD-1 expressions, concentration of cytokine, and ribonucleic acid sequencing (seq)/T-cell receptor seq etc. will be monitored. The measurements of biomarkers in changes over time from baseline to several time-points will be performed by using generalized linear mixed effects modeling with a Benjamini-Hochberg correction to control for false discovery rates.
Time Frame: Baseline up to 3 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Biomarkers or Serial Measurements of Biomarkers Associated With Survival Outcomes
Description: The Kaplan-Meier method and log-rank test will be used to estimate the distribution of survival between/among different marker strata. Univariate or Multivariate cox proportional hazard models will be employed to explore the significance of biomarkers on survival outcomes, while adjusting for the potential prognostic factors. The interaction effects between treatment and biomarkers also will be evaluated. Serial measurements of biomarkers will be estimated at baseline, end of induction, post-cycle 1, 2, 4, and 6, every 3 months during maintenance, one year, and end of treatment when applicable. Landmark analysis or joint modeling will be used to assess serial measurements of biomarkers dynamical impacts on survival outcomes, where appropriate.
Time Frame: Baseline up to 3 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Biomarkers Effects Between Treatment Arms
Description: The associations between treatment arms and baseline biomarkers will be evaluated using Chi-squared test/ Fisher's exact test, analysis of variance and the Mann-Whitney U tests as appropriate. Trajectory trends of the changes in markers' values or status across the measurement time will be explored using generalized linear mixed models. The bar plots and trajectory time plots will visually show the differences over time between treatment arms. The associations between markers and the demographic/prognostic factors will also be assessed using the similar statistical methods.
Time Frame: Up to 3 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Correlations Between Biomarkers
Description: The correlations between biomarkers will be evaluated using Pearson/Spearman rank-order correlation coefficients, Chi-squared/Fisher's exact tests, and Wilcoxon rank sun / Kruskal-Wallis tests as appropriate. A scatter plot, boxplot, and mosaic plot will also be generated for visualization. The multiplicity of the endpoints will be adjusted using the correction of Benjamini and Hochberg.
Time Frame: Up to 3 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: MRD Assessment
Description: Library preparation, sequencing, and analysis will be performed with TwinStrand's optimized workflow, and TwinStrand's bioinformatics core will perform all analyses related to assay output.
Time Frame: Up to 3 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Cytokine Panel Analysis
Description: IFN-gamma+/CD3+/ CD4+ or IFN-gamma+/CD3+/CD8+ events will be gated and percentages of the total CD4+ and CD8+ T cells will be determined. Will compare levels of leukemia specific T-cell.
Time Frame: At day 30 (after administration of pembrolizumab and count recovery) and after cycles 2, 4, and 6 (each cycle is 28 days)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Expression of PD-1, PD-L1 in Acute Myeloid Leukemia (AML) Bone Marrow (BM)
Description: An association of clinical response with the expression of PD-L1 AML BM cells will be assessed by a Pearson chi-square test on a 2x2 table of frequencies.
Time Frame: At day 14 and at time of count recovery
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Dynamic Change of Immune Subsets
Description: Statistical analyses of the frequency of CD8+, CD4+, Foxp3 regulatory T cells, CD8+/Foxp3+ Tregs, central memory T cell/effector memory T cell re-expressed CD45RA (TEMRA), effector memory T cell/TEMRA, the percentage of Ki67 and GzmB in PD-1+, Eomes+ CD8 T cells to compare changes over time from baseline to several time-points will be performed by using mixed effects modeling with a Benjamini-Hochberg correction to control for false discovery rates.
Time Frame: Baseline up to cycle 6 (each cycle is 28 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Arm I (AZA, VEN) | Arm II (AZA, VEN, Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 18/29 | 22/29
Serious Adverse Events (participants affected / at risk) | 28/29 | 29/29
Other Adverse Events (participants affected / at risk) | 26/29 | 26/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (AZA, VEN) (N=29) | Arm II (AZA, VEN, Pembrolizumab) (N=29)
Anemia (Blood and lymphatic system disorders) | 11 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0
Death NOS (General disorders) | 1 | 1
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 2
Fever (General disorders) | 0 | 1
General and admin site - Other - Volume overload (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 1
GI disorders - Other, specify - Diverticular abscess (Gastrointestinal disorders) | 0 | 2
GI disorders - Other, specify - Diverticulitis (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Hepatobiliary disorders - Other - Choledocholithiasis (Hepatobiliary disorders) | 0 | 1
Infections & infestations - Other - COVID 19 Infection (Infections and infestations) | 0 | 0
Infections & infestations - Other - Sepsis (Infections and infestations) | 1 | 7
Lung infection (Infections and infestations) | 3 | 1
Pelvic infection (Infections and infestations) | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 2 | 2
Skin infection (Infections and infestations) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 4
ALT increased (Investigations) | 0 | 4
AST increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Cardiac troponin I increased (Investigations) | 0 | 0
EKG QT corrected interval prolong (Investigations) | 1 | 1
Fibrinogen decreased (Investigations) | 0 | 18
Lymphocyte count decreased (Investigations) | 14 | 21
Neutrophil count decreased (Investigations) | 19 | 19
Platelet count decreased (Investigations) | 15 | 0
Weight loss (Investigations) | 1 | 24
White blood cell decreased (Investigations) | 24 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0
Musculoskel/connect tissue -Other - Knee effusion (hemarthrosis) (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neoplasms - Other - AML disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasms - Other - AML progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasms - Other - peripheral blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 0 | 4
Syncope (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0
Genital edema (Reproductive system and breast disorders) | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Resp, thoracic & mediast - Other - Lung Nodules (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0
Surgical and medical - Other - knee ablation (Surgical and medical procedures) | 1 | 1
Hematoma (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 5
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (AZA, VEN) (N=29) | Arm II (AZA, VEN, Pembrolizumab) (N=29)
Anemia (Blood and lymphatic system disorders) | 16 | 20
Blood/Lymph - Other - idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Blood/Lymph - Other - Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Blood/Lymph - Other - Thryoiditis (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 10
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 4
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac disorders - Other - Coronary Artery Disease (Cardiac disorders) | 0 | 1
Cardiac disorders - Other - Murmur (Cardiac disorders) | 1 | 0
Cardiac disorders - Other - tachycardia nos (Cardiac disorders) | 0 | 1
Cardiac disorders - Other - tachycardia NOS (Cardiac disorders) | 1 | 0
Heart failure (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 6 | 2
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Ear and Labyrinth - Other - ear fullness (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Endocrine disorders - Other - Euthyroid Sick Syndrome (Endocrine disorders) | 0 | 1
Endocrine disorders - Other - Hypervolemia (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1
Blurred vision (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 2
Eye disorders - Other, specify - Blepharitis (Eye disorders) | 0 | 1
Eye disorders - Other, specify - Bloodshot eyes / minor hemorrhage (Eye disorders) | 1 | 0
Eye disorders - Other, specify - conjuctivitis (Eye disorders) | 0 | 1
Eye disorders - Other, specify - erythema of left eye (Eye disorders) | 0 | 1
Eye disorders - Other, specify - pruritus of left eye (Eye disorders) | 0 | 1
Eye disorders - Other, specify - Rt Eye Stye (Eye disorders) | 1 | 0
Eye disorders - Other, specify - superficial punctuate epithelial erosions bilateral eyes (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 0 | 1
Floaters (Eye disorders) | 0 | 1
Retinal vascular disorder (Eye disorders) | 1 | 0
Scleral disorder (Eye disorders) | 1 | 0
Chills (General disorders) | 4 | 5
Edema face (General disorders) | 0 | 1
Edema limbs (General disorders) | 5 | 11
Fatigue (General disorders) | 10 | 12
Fever (General disorders) | 5 | 8
General and admin site - Other - bilateral forearm flaking (General disorders) | 0 | 1
General and admin site - Other - bilateral forearm redness (General disorders) | 0 | 1
General and admin site - Other - Gum Pain (General disorders) | 0 | 1
General and admin site - Other - temperature increased (General disorders) | 1 | 0
General and admin site - Other - vaccine reaction (General disorders) | 0 | 1
Generalized edema (General disorders) | 2 | 3
Injection site reaction (General disorders) | 2 | 2
Malaise (General disorders) | 1 | 1
Neck edema (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 3
Pain (General disorders) | 2 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Anal fissure (Gastrointestinal disorders) | 0 | 1
Anal pain (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 14 | 17
Diarrhea (Gastrointestinal disorders) | 12 | 14
Dry mouth (Gastrointestinal disorders) | 2 | 3
Dysphagia (Gastrointestinal disorders) | 2 | 3
Esophagitis (Gastrointestinal disorders) | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 1
GI disorders - Other, specify - blood in stool (Gastrointestinal disorders) | 0 | 1
GI disorders - Other, specify - Diverticulitis (Gastrointestinal disorders) | 0 | 2
GI disorders - Other, specify - Early Satiety (Gastrointestinal disorders) | 0 | 1
GI disorders - Other, specify - GI Bleed (Gastrointestinal disorders) | 1 | 0
GI disorders - Other, specify - left lip lesion NOS (Gastrointestinal disorders) | 1 | 0
GI disorders - Other, specify - malnutrition (Gastrointestinal disorders) | 1 | 0
GI disorders - Other, specify - melena (Gastrointestinal disorders) | 1 | 1
GI disorders - Other, specify - pancreatic lesions (Gastrointestinal disorders) | 1 | 0
GI disorders - Other, specify - tenesmus (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 3
Mucositis oral (Gastrointestinal disorders) | 7 | 3
Nausea (Gastrointestinal disorders) | 16 | 10
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 2
Rectal pain (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 3
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 7 | 6
Hepatobiliary disorders - Other - liver cirrhosis (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 2 | 2
Appendicitis (Infections and infestations) | 0 | 1
Bacteremia (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Infections & infestations - Other - bladder (Infections and infestations) | 1 | 0
Infections & infestations - Other - C.difficile infection (Infections and infestations) | 0 | 1
Infections & infestations - Other - COVID-19 (Infections and infestations) | 1 | 0
Infections & infestations - Other - COVID-19 infection (Infections and infestations) | 1 | 0
Infections & infestations - Other - COVID19 infection (Infections and infestations) | 1 | 0
Infections & infestations - Other - osteomyelitis (Infections and infestations) | 1 | 0
Infections & infestations - Other - Sepsis (Infections and infestations) | 1 | 0
Infections & infestations - Other - Whooping cough (pertussis) (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 3 | 4
Pharyngitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 3
Small intestine infection (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 2 | 1
Wound infection (Infections and infestations) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 5 | 1
Fall (Injury, poisoning and procedural complications) | 6 | 2
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Injury/poison/procedure - Other - abrasion of bilateral knees (Injury, poisoning and procedural complications) | 0 | 1
Injury/poison/procedure - Other - abrasion of left elbow (Injury, poisoning and procedural complications) | 0 | 1
Injury/poison/procedure - Other - abrasion to left eye (Injury, poisoning and procedural complications) | 0 | 1
Injury/poison/procedure - Other - abrasion to left knee (Injury, poisoning and procedural complications) | 0 | 1
Injury/poison/procedure - Other - laceration of left forehead (Injury, poisoning and procedural complications) | 0 | 1
Injury/poison/procedure - Other - left hip injury (Injury, poisoning and procedural complications) | 0 | 1
Injury/poison/procedure - Other - pain at r. hohn (Injury, poisoning and procedural complications) | 0 | 1
Injury/poison/procedure - Other - r. ankle sprain (Injury, poisoning and procedural complications) | 0 | 1
Injury/poison/procedure - Other - skin tear (Injury, poisoning and procedural complications) | 1 | 0
Injury/poison/procedure - Other - to left wrist (Injury, poisoning and procedural complications) | 1 | 0
Injury/poison/procedure - Other - VAD site bleeding (Injury, poisoning and procedural complications) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 4
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Activated PTT prolonged (Investigations) | 1 | 2
Alkaline phosphatase increased (Investigations) | 5 | 8
ALT increased (Investigations) | 4 | 9
AST increased (Investigations) | 5 | 10
Blood bicarbonate decreased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 11 | 8
Cardiac troponin I increased (Investigations) | 0 | 1
Cardiac troponin T increased (Investigations) | 0 | 1
Creatinine increased (Investigations) | 6 | 9
EKG QT corrected interval prolong (Investigations) | 2 | 2
Elevated LDH (Investigations) | 2 | 4
Elevated TSH (Investigations) | 0 | 2
Fibrinogen decreased (Investigations) | 0 | 1
INR increased (Investigations) | 4 | 8
Investigations - Other, specify - CRP increased (Investigations) | 0 | 1
Investigations - Other, specify - D-Dimer, Quantified Increased (Investigations) | 1 | 0
Investigations - Other, specify - Fibrinogen increased (Investigations) | 1 | 0
Investigations - Other, specify - Monocyte count decreased (Investigations) | 1 | 0
Investigations - Other, specify - vitamin d deficiency (Investigations) | 1 | 0
Investigations - Other, specify - WBC increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 18 | 21
Neutrophil count decreased (Investigations) | 20 | 21
Platelet count decreased (Investigations) | 20 | 24
Weight loss (Investigations) | 2 | 6
White blood cell decreased (Investigations) | 25 | 24
Anorexia (Metabolism and nutrition disorders) | 7 | 10
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 11
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 3
Hyperphosphatemia (Metabolism and nutrition disorders) | 3 | 6
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 | 16
Hypocalcemia (Metabolism and nutrition disorders) | 10 | 12
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 9 | 16
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 5
Hyponatremia (Metabolism and nutrition disorders) | 9 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 7 | 8
Metabolism and nutrition - Other - Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Metabolism and nutrition - Other - Uric acid decreased (Metabolism and nutrition disorders) | 1 | 0
Metabolism and nutrition - Other - Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskel/connect tissue -Other - Bilateral Leg Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskel/connect tissue -Other - degenerative disc disease (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskel/connect tissue -Other - gout flare up (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskel/connect tissue -Other - groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskel/connect tissue -Other - hip soreness in the mornings and when standing (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskel/connect tissue -Other - Iliac bone sclerosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskel/connect tissue -Other - Knee effusion (hemarthrosis) (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskel/connect tissue -Other - Knee effusion (recurrent) (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskel/connect tissue -Other - disease of cervical and lumbar spine (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskel/connect tissue -Other - pain at bone marrow biopsy site (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskel/connect tissue -Other - sclerotic lesions (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskel/connect tissue -Other - Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskel/connect tissue -Other - subcutaneous soft mass r upper quadrant (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 6
Rotator cuff injury (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms - Other - Bakers Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasms - Other - breast mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasms - Other - complex baker's cyst - Right knee (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasms - Other - peripheral blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasms - Other - Precancerous skin lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasms - Other - thyroid nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 1
Concentration impairment (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 5 | 6
Dysgeusia (Nervous system disorders) | 1 | 6
Headache (Nervous system disorders) | 5 | 6
Lethargy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 2
Nervous system - Other - benzodiazapine withdrawal (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 2 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 2 | 3
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 0
Confusion (Psychiatric disorders) | 0 | 3
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Hallucinations (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 6 | 3
Psychiatric disorders - Other - parasomnia, night terror (Psychiatric disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 4
Dysuria (Renal and urinary disorders) | 4 | 2
Glucosuria (Renal and urinary disorders) | 2 | 2
Hematuria (Renal and urinary disorders) | 3 | 6
Proteinuria (Renal and urinary disorders) | 1 | 4
Renal & urinary disorders - Other - eGFR decreased (Renal and urinary disorders) | 1 | 0
Renal calculi (Renal and urinary disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 2 | 4
Urinary incontinence (Renal and urinary disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 1 | 3
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 2 | 0
Urine discoloration (Renal and urinary disorders) | 1 | 3
Genital edema (Reproductive system and breast disorders) | 1 | 0
Testicular disorder (Reproductive system and breast disorders) | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Resp, thoracic & mediast - Other - hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Resp, thoracic & mediast - Other - incidental lung nodules (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Resp, thoracic & mediast - Other - Pulmonary nodule (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 5
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 6
Skin & subcutaneous tissue -Other - erythema at CVC of r. jugular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin & subcutaneous tissue -Other - Erythematous Petechial Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin & subcutaneous tissue -Other - petechia (Skin and subcutaneous tissue disorders) | 1 | 0
Skin & subcutaneous tissue -Other - petechial non-pruritic rash of bilateral feet (Skin and subcutaneous tissue disorders) | 1 | 0
Skin & subcutaneous tissue -Other - r. femoral hernia (Skin and subcutaneous tissue disorders) | 0 | 1
Skin & subcutaneous tissue -Other - rash of back (Skin and subcutaneous tissue disorders) | 1 | 0
Skin & subcutaneous tissue -Other - rash of neck NOS (Skin and subcutaneous tissue disorders) | 0 | 1
Skin & subcutaneous tissue -Other - rash of r. ankle NOS (Skin and subcutaneous tissue disorders) | 0 | 1
Skin & subcutaneous tissue -Other - redness and draining at PICC site (Skin and subcutaneous tissue disorders) | 1 | 0
Skin & subcutaneous tissue -Other - Scattered petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Skin & subcutaneous tissue -Other - skin abrasion ( r. Knee) (Skin and subcutaneous tissue disorders) | 1 | 0
Skin & subcutaneous tissue -Other - sunburn of nose (Skin and subcutaneous tissue disorders) | 0 | 1
Skin & subcutaneous tissue -Other - Sweet Syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Skin & subcutaneous tissue -Other - Sweet's syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Skin & subcutaneous tissue -Other - wound to l. buttock NOS (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Surgical and medical - Other - PICC placement (Surgical and medical procedures) | 0 | 1
Hematoma (Vascular disorders) | 2 | 3
Hot flashes (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 4 | 5
Hypotension (Vascular disorders) | 8 | 8
Thromboembolic event (Vascular disorders) | 3 | 1
Vascular disorders - Other - orthostatic hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT04284787/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT04284787/ICF_001.pdf